CLINICAL TRIAL: NCT03233009
Title: A Human Subject 24 Hour Patch Test to Assess the Irritation Potential of Four Skin Serum Products
Brief Title: To Investigate Primary Irritation Potential of Four Skin Serum Products on Human Subjects Assessed by 24 Hour Patch Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 207235
Record Dates: First submitted 2017-07-07; First posted 2017-07-28 (Actual); Results first posted 2018-09-07 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-12

CONDITIONS: Skin Care
MeSH Terms: interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Test Product 1 (Experimental): Participants will topically apply test product 1 via semi occlusive patch.
  Interventions: Other: Experimental Daily Defense Serum A
- Test Product 2 (Experimental): Participants will topically apply test product 2 via semi occlusive patch.
  Interventions: Other: Experimental Daily Defense Serum C
- Test Product 3 (Experimental): Participants will topically apply test product 3 via semi occlusive patch.
  Interventions: Other: Experimental Daily Defense Serum G
- Test Product 4 (Experimental): Participants will topically apply test product 4 via semi occlusive patch.
  Interventions: Other: Experimental Daily Defense Serum N
- Reference Product (Sham Comparator): Participants will topically apply Reference product via semi occlusive patch.
  Interventions: Other: Saline Solution Sodium Chloride

INTERVENTIONS:
Other: Experimental Daily Defense Serum A — Participants will apply 0.02mL/cm2 of product topically via semi-occlusive patches onto dorsum (Scapular region).
  Arms: Test Product 1
Other: Experimental Daily Defense Serum C — Participants will apply 0.02mL/cm2 of product topically via semi-occlusive patches onto dorsum (Scapular region).
  Arms: Test Product 2
Other: Experimental Daily Defense Serum G — Participants will apply 0.02mL/cm2 of product topically via semi-occlusive patches onto dorsum (Scapular region).
  Arms: Test Product 3
Other: Experimental Daily Defense Serum N — Participants will apply 0.02mL/cm2 of product topically via semi-occlusive patches onto dorsum (Scapular region).
  Arms: Test Product 4
Other: Saline Solution Sodium Chloride — Participants will apply 0.02mL/cm2 of product topically via semi-occlusive patches onto dorsum (Scapular region).
  Arms: Reference Product

SUMMARY:
To assess the irritation potential of four prototype daily defense serum formulations after 24 (± 2) hours under semi-occlusive patch application to the skin of healthy volunteers.

DETAILED DESCRIPTION:
This is an evaluator (single) blind, test site randomized and intra-subject comparison patch test study to evaluate the cutaneous irritation potential of four experimental daily defense serum formulations, including a saline solution as a negative control.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* General health: Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination and participants must have intact skin on the proposed application site; dorsum (scapular region).
* Fitzpatrick photo type I to IV.
* Agreement to comply with the procedures and requirements of the study and to attend the scheduled assessment visits.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* Any history of significant dermatological diseases or conditions or medical conditions known to alter skin appearance or physiologic response (e.g. diabetes,) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction.
* Presence of open sores, pimples, or cysts at the application site.
* Active dermatosis (local or disseminated) that might interfere with the results of the study
* Considered immune compromised.
* History of diseases aggravated or triggered by ultraviolet radiation.
* Participants with dermatographism.
* Currently using any medication which in the opinion of the investigator, may affect the evaluation of the study product, or place the participant at undue risk.
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs, and corticosteroids up to 2 weeks before Screening visit.
* Oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit.
* Intention of being vaccinated during the study period or vaccination within 3 weeks of the Screening visit.
* Currently receiving allergy injections, or due to receive an injection within 7 days prior to Visit 1, or expects to begin injections during study participation.
* Previous history of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, cosmetics or medication.
* Known or suspected intolerance or hypersensitivity to any of the study materials (or closely related compounds) or any of their stated ingredients, including any component of the patches.
* History of sensitization in a previous patch study.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the Screening visit.
* Previous participation in this study.
* Recent history (within the last 5 years) of alcohol or other substance abuse.
* Intense sunlight exposure or sun tanning sessions up to 30 days before the Screening evaluation Intention of bathing, sauna, water sports, or activities that lead to intense sweating.
* Any participant who, in the judgment of the Investigator, should not participate in the study.
* Any skin marks on the test site that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, vascular malformations, scars, tattoos, excessive hair, numerous freckles).
* Prisoner or involuntary incarcerated participant.
* Participant from an indigenous tribe.
* An employee of the sponsor or the study site or members of their immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Valinhos, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=207235&attachmentIdentifier=86ec8b21-ef92-4a57-9623-7afe670832a7&fileName=gsk-207235-clinical-study-report-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were enrolled at one center in Brazil.
Pre-assignment Details: A total of 46 participants were screened, out of which 3 participants did not meet study criteria, 43 participants were enrolled in the study out of which 3 participants withdrew their consent. Remaining 40 participants were randomized to the study.
Groups:
- Overall Participants: All participants enrolled in the study received all the study products. Test and control products were applied to a paper disc (or cell) contained within an adhesive patch in a randomized manner. The number of cells available on the patch test tape is 6 (but only 5 cells were used, 4 test and 1 reference products). The patch was then applied onto the dorsum (scapula region) of each participant for a period of 24 ± 2 hours, the sequence of the product application to the cells was as per the randomization schedule.
Period: Overall Study
Arm/Group | Overall Participants
Started | 40
Test Product 1 | 39
Test Product 2 | 39
Test Product 3 | 39
Test Product 4 | 39
Reference Product | 39
Completed (1 participant lost to follow-up was removed from all the treatment arms.) | 39
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline population reflects the safety population. The safety population (N= 40) included all participants who received any of the test products
Groups:
- Overall Participants: All participants randomized to the study. Test and control products were applied to a paper disc (or cell) contained within an adhesive patch. The number of cells available on the patch test tape is 6 (but only 5 cells were used, 4 test and 1 reference products). The patch was then applied onto the dorsum (scapula region) of each participant for a period of 24 ± 2 hours, the sequence of the product application to the cells was as per the randomization schedule.
Arm/Group | Overall Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Dermal Response Score at 15-30 Minutes Post Patch Removal
Description: Product tolerability was assessed by Dermal Response Score. Test sites were evaluated 15-30 minutes following patch removal on Day 2 post 24 hrs of patch application. Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test site.
Time Frame: At Day 2 (15-30 minutes post patch removal)
Population: The ITT (N= 39) population included all participants who were randomized into the study and have skin irritation scores from at least one of the test sites available.
Measure: Count of Participants; unit: Participants
Groups:
- Test Product 1: This arm includes data from the test sites where test product 1 was applied.
- Test Product 2: This arm includes data from the test sites where test product 2 was applied.
- Test Product 3: This arm includes data from the test sites where test product 3 was applied.
- Test Product 4: This arm includes data from the test sites where test product 4 was applied.
- Reference Product: This arm includes data from the test sites where reference product was applied.
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference Product
Number analyzed (Participants) | 39 | 39 | 39 | 39 | 39
Participants
  Missing | 0 | 0 | 0 | 0 | 0
  0 | 39 | 39 | 39 | 39 | 39
  1 | 0 | 0 | 0 | 0 | 0
  2 | 0 | 0 | 0 | 0 | 0
  3 | 0 | 0 | 0 | 0 | 0
  4 | 0 | 0 | 0 | 0 | 0
  5 | 0 | 0 | 0 | 0 | 0
  6 | 0 | 0 | 0 | 0 | 0
  7 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Frequency of Dermal Response Score at 24 Hours Post Patch Removal
Description: Product tolerability was assessed by Dermal Response Score. Test sites were evaluated 24 hours following patch removal on Day 3 post 48 hrs of patch application. Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test site.
Time Frame: At Day 3 (24 hours post patch removal)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference Product
Number analyzed (Participants) | 39 | 39 | 39 | 39 | 39
Participants
  Missing | 0 | 0 | 0 | 0 | 0
  0 | 39 | 39 | 39 | 39 | 39
  1 | 0 | 0 | 0 | 0 | 0
  2 | 0 | 0 | 0 | 0 | 0
  3 | 0 | 0 | 0 | 0 | 0
  4 | 0 | 0 | 0 | 0 | 0
  5 | 0 | 0 | 0 | 0 | 0
  6 | 0 | 0 | 0 | 0 | 0
  7 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Frequency of Dermal Response Score at 48 Hours Post Patch Removal
Description: Product tolerability was assessed by Dermal Response Score. Test sites were evaluated 48 hours following patch removal on Day 4 post 72 hours of patch application. Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test site.
Time Frame: At Day 4 (48 hours post patch removal)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference Product
Number analyzed (Participants) | 39 | 39 | 39 | 39 | 39
Participants
  Missing | 0 | 0 | 0 | 0 | 0
  0 | 39 | 39 | 39 | 39 | 39
  1 | 0 | 0 | 0 | 0 | 0
  2 | 0 | 0 | 0 | 0 | 0
  3 | 0 | 0 | 0 | 0 | 0
  4 | 0 | 0 | 0 | 0 | 0
  5 | 0 | 0 | 0 | 0 | 0
  6 | 0 | 0 | 0 | 0 | 0
  7 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Average Dermal Response Score at 30 Minutes Post Patch Removal
Description: Product tolerability was assessed by Dermal Response Score. Test sites were evaluated 15-30 minutes following patch removal on Day 2 post 24 hours of patch application. Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test site.
Time Frame: At Day 2 (15-30 minutes post patch removal)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference Product
Number analyzed (Participants) | 39 | 39 | 39 | 39 | 39
Score on Scale | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

5. Primary Outcome: Average Dermal Response Score at 24 Hours Post Patch Removal
Description: Product tolerability was assessed by Dermal Response Score. Test sites were evaluated 24 hours following patch removal on Day 3 post 48 hours of patch application. Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test site.
Time Frame: At Day 3 (24 hours post patch removal)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference Product
Number analyzed (Participants) | 39 | 39 | 39 | 39 | 39
Score on Scale | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

6. Primary Outcome: Average Dermal Response Score at 48 Hours Post Patch Removal
Description: as for outcome 3
Time Frame: At Day 4 (48 hours post patch removal)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference Product
Number analyzed (Participants) | 39 | 39 | 39 | 39 | 39
Score on scale | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

7. Secondary Outcome: Number of Participants With Combined Skin Irritation (Dermal Response) Scores at 30 Minutes, 24 Hours and 48 Hours Post Patch Removal
Description: A trained assessor assessed all patch sites.Following scores were used to express response observed at time of examination:0=No evidence of irritation,1=Minimal erythema;barely perceptible,2=Definite erythema,readily visible;or minimal edema; or minimal papular response,3=Erythema and papules,4=Definite edema,5=Erythema, edema,and papules,6=Vesicular eruption,7=Strong reaction spreading beyond test site.Other features indicative irritation (Superficial irritation) scores were:GradeA/Score0=Slight glazed appearance,GradeB/Score1=Marked glazing,GradeC/Score2=Glazing with peeling and cracking,GradeF/Score3=Glazing with fissures,Grade G/Score 3=Film of dried serous exudate covering all or portion of patch,Grade H/Score3=Small petechial erosions and/or scabs.The letter grades were converted to scores.Superficial irritation scores were only provided if there was a dermal response score >0.No effect is 0 score(i.e. no evidence).Full Range 0-10.Lower score indicates better product tolerabily
Time Frame: At Day 2 (15-30 minutes), Day 3 (24 hours) and Day 4 (48 hours) post patch removal
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference Product
Number analyzed (Participants) | 39 | 39 | 39 | 39 | 39
Participants
  Day 2 (15-30 minutes): No effect | 39 | 39 | 39 | 39 | 39
  Day 2 (15-30 minutes): Missing | 0 | 0 | 0 | 0 | 0
  Day 2 (15-30 minutes): Grade A/Score 0 | 0 | 0 | 0 | 0 | 0
  Day 2 (15-30 minutes): Grade B/Score 1 | 0 | 0 | 0 | 0 | 0
  Day 2 (15-30 minutes): Grade C/Score 2 | 0 | 0 | 0 | 0 | 0
  Day 2 (15-30 minutes): Grade F/Score 3 | 0 | 0 | 0 | 0 | 0
  Day 2 (15-30 minutes): Grade G/Score 3 | 0 | 0 | 0 | 0 | 0
  Day 2 (15-30 minutes): Grade H/Score 3 | 0 | 0 | 0 | 0 | 0
  Day 3 (24 hours): No effect | 39 | 39 | 39 | 39 | 39
  Day 3 (24 hours): Missing | 0 | 0 | 0 | 0 | 0
  Day 3 (24 hours): Grade A/Score 0 | 0 | 0 | 0 | 0 | 0
  Day 3 (24 hours): Grade B/Score 1 | 0 | 0 | 0 | 0 | 0
  Day 3 (24 hours): Grade C/Score 2 | 0 | 0 | 0 | 0 | 0
  Day 3 (24 hours): Grade F/Score 3 | 0 | 0 | 0 | 0 | 0
  Day 3 (24 hours): Grade G/Score 3 | 0 | 0 | 0 | 0 | 0
  Day 3 (24 hours): Grade H/Score 3 | 0 | 0 | 0 | 0 | 0
  Day 4 (48 hours): No effect | 39 | 39 | 39 | 39 | 39
  Day 4 (48 hours): Missing | 0 | 0 | 0 | 0 | 0
  Day 4 (48 hours): Grade A/Score 0 | 0 | 0 | 0 | 0 | 0
  Day 4 (48 hours): Grade B/Score 1 | 0 | 0 | 0 | 0 | 0
  Day 4 (48 hours): Grade C/Score 2 | 0 | 0 | 0 | 0 | 0
  Day 4 (48 hours): Grade F/Score 3 | 0 | 0 | 0 | 0 | 0
  Day 4 (48 hours): Grade G/Score 3 | 0 | 0 | 0 | 0 | 0
  Day 4 (48 hours): Grade H/Score 3 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 4 days
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Test Product 4 | Reference Product | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT03233009/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT03233009/SAP_001.pdf